CLINICAL TRIAL: NCT00374452
Title: VISN Collaborative for Improving Hypertension Management With ATHENA-HTN
Acronym: HTN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IMV 04-062
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Hypertension
Keywords: hypertension; practice guidelines; quality of health care; decision support systems; evidence-based medicine; medical informatics
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATHENA-CDS-HTN plus Guideline Link (Experimental): ATHENA-CDS-HTN plus Guideline Link. ATHENA-CDS-HTN display on the cover sheet of electronic health record, plus link to the guidelines
  Interventions: Other: ATHENA-CDS-HTN plus Guideline Link
- Guideline Link Only (Other): Guideline Link Only. Link to The Seventh Report of the Joint National Committee on Prevention Detection and Treatment of High Blood Pressure (JNC7) and to VA-Department of Defense (DoD) hypertension guidelines
  Interventions: Other: Guideline Link Only

INTERVENTIONS:
Other: ATHENA-CDS-HTN plus Guideline Link — ATHENA display provides guideline-based recommendations to clinicians at the time of patient care.
  Arms: ATHENA-CDS-HTN plus Guideline Link
Other: Guideline Link Only — Primary care providers were sent, once, a link (URL) to the VA/DoD and JNC7 hypertension guidelines.
  Arms: Guideline Link Only

SUMMARY:
This project is a VA HSR&D-funded Quality Enhancement Research Initiative (QUERI) project to translate into practice evidence about clinical management of primary hypertension. The project aims to contribute to quality improvement of care for patients with primary hypertension. The project implemented a clinical decision support (CDS) system for primary care clinicians and evaluated the implementation by studying the following: impact on the clinicians' prescribing and their patients' blood pressures; the clinician satisfaction with the CDS; and organizational factors in the implementation.

DETAILED DESCRIPTION:
Background / Rationale:

Despite the existence of evidence-based guidelines, there is a gap between evidence-based recommended best medical practice and actual practice. In previous work, we used hypertension as a model to study the translation of research regarding clinical blood pressure targets and drug choice into primary care practice through computer-based implementation of clinical practice guidelines. In collaboration with experts in guideline-automation at Stanford Center for Biomedical Informatics Research (BMIR) (formerly known as Stanford Medical Informatics, SMI), we developed an innovative clinical decision support system: ATHENA-CDS-HTN (hypertension) also known as ATHENA-HTN. ATHENA-HTN is a knowledge-based CDS that uses knowledge bases (KBs) of clinical knowledge of hypertension encoded into computable formats. Clinical data from an electronic health records system is processed with the knowledge in the KB by an execution engine (also known as a guideline interpreter) that generates patient-specific outputs with conclusions about the current state of the patient with respect to the guidelines as shown in the patient's electronic health record data and also generates detailed recommendations for next steps in clinical management of the patient's hypertension. The system is designed to take account of multiple data elements in the patients' clinical data including co-morbid diagnoses that are relevant to hypertension and its treatment, other medications currently prescribed, history of adverse drug reactions/events, and selected laboratory values relevant to hypertension and its management. In previous work, we had demonstrated that deploying this CDS system in VA primary care clinics was feasible and that clinicians found the system usable and useful, as shown by their actual extensive use of the system and their response to a questionnaire survey. The current project was funded by the Department of Veterans Affairs Health Services Research and Development (HSR&D), under a special funding initiative for Quality Enhancement Initiative (QUERI) projects designed to improve care for hypertension by collaboration with a Veterans Integrated Service Network (VISN) to implement programs to encourage use of established best-practices for managing hypertension according to evidence-based guidelines available at the time of the study. These studies were known as "VISN Collaboratives". The studies did not involve any new drugs or new uses of established drugs, but rather encouraging use of established drugs recommended in standard evidence-based guidelines for care. The focus of the study was implementation of existing known best practices in managing hypertension, using the CDS as a vehicle to bring information to the point-of-care, with detailed individualized recommendations about patients presented to the primary care provider at the time the provider sees patients in scheduled outpatient primary care clinic visits.

Objective(s):

Our objectives in this VISN Implementation Collaborative included: (1) implement evidence-based guidelines for hypertension in a CDS system by upgrading the ATHENA-HTN knowledge-base (KB) to the most recent guidelines; (2) deploy the CDS system in 5 medical centers within VISN 1 to generate individualized recommendations to primary care clinicians caring for patients in outpatient clinics; (3) evaluate the implementation including the organizational aspects.

Methods:

In Phase 1 we plan to update the KB and conduct offline testing; to revise the M (formerly known as MUMPS) program that extracts patient data daily from VistA to extract additional data elements; to streamline the system architecture to make it easier to implement in multiple sites; to work with the site-PIs to obtain IRB approval at 5 implementation sites in VISN 1 plus the coordinating site at VA Palo Alto; to improve the user interface design; to identify and resolve issues in implementing new information technology in multiple different VA medical centers (VAMC) with different Computerized Patient Record System (CPRS) implementations and different methods of distributing computer access to clinicians; to train the site PIs in use of the system; and perform baseline data analysis to inform the randomization. In Phase 2 we plan to recruit primary care providers from the participating 5 medical centers in VISN 1; randomize clinics to ATHENA-HTN intervention or usual care; deploy the system for intervention providers; train intervention providers in use of the system; and conduct a 12-month clinical trial of the system.

Status:

The project has been completed. We completed Institutional Review Board (IRB) approvals at all five medical centers. We updated the knowledge base of computable knowledge regarding hypertension and conducted offline testing. Our system was deployed to all five medical centers. While we were preparing for deployment of the CDS, one site changed from a rich-client environment to a thin-client environment for the medical center computers; we developed new code to run the system in a thin client environment. The previous programming computed recommendations of the CDS based on clinical data available the night before the clinic visit (in order to pre-compute advisories for faster display during clinic); in this project we developed software code to obtain automatic blood pressure updates for the day of visit if these were entered by clinical staff at the time of the visit. VA Palo Alto staff worked with staff at each VAMC to validate clinical data extraction at each site. We developed code for a clinician to select, optionally, for blood pressure write-back to VA VistA so that if clinicians entered to our CDS a blood pressure measurement that they had just taken so they could view updated recommendations based on the repeat blood pressure they would not also have to enter that blood pressure separately to electronic health record. We recruited primary care providers (clinicians) at each of 5 medical centers to participate in the project. One of the 5 medical centers completed the installation of the ATHENA-HTN system, but did not continue with the intervention period, so the intervention included 4 rather than 5 medical centers. Our site-principal investigators and project coordinator trained intervention providers on use of the system by offering short phone calls for training or in-person introduction, and by making the system available for a short period of time for familiarity. Records of patients seen by the clinicians in this training period were excluded from analyses. We completed a 6-8 month intervention period for the clinical trial at the 4 participating medical centers. Our random allocation was at clinic level, where a clinic is a substation of a medical center (station). Before initiating data analyses, we prepared a detailed data analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* Must be primary care clinicians (for example, physician or nurse practitioner) at one of the participating VA medical centers. This study is NOT recruiting patients.
* The primary care clinician must have a panel of patients for whom he or she provides direct care.

Exclusion Criteria:

* Anyone who does not meet inclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-01; Primary Completion 2010-05 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary K. Goldstein, MD MS, Principal Investigator — VA Palo Alto Health Care System
Locations (7):
- United States (7):
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA Connecticut Health Care System (Newington), Newington, Connecticut
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, Bedford, Massachusetts
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Medical Center, Manchester, Manchester, New Hampshire
  - VA Medical Center, Providence, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martins SB, Lai S, Tu S, Shankar R, Hastings SN, Hoffman BB, Dipilla N, Goldstein MK. Offline testing of the ATHENA Hypertension decision support system knowledge base to improve the accuracy of recommendations. AMIA Annu Symp Proc. 2006;2006:539-43. PMID 17238399
- [Result] Chan AS, Shankar RD, Coleman RW, Matins SB, Hoffman BB, Goldstein MK. Leveraging point-of-care clinician feedback to study barriers to guideline adherence. AMIA Annu Symp Proc. 2005;2005:915. PMID 16779202
- [Result] Trafton J, Martins S, Michel M, Lewis E, Wang D, Combs A, Scates N, Tu S, Goldstein MK. Evaluation of the acceptability and usability of a decision support system to encourage safe and effective use of opioid therapy for chronic, noncancer pain by primary care providers. Pain Med. 2010 Apr;11(4):575-85. doi: 10.1111/j.1526-4637.2010.00818.x. Epub 2010 Mar 1. PMID 20202142
- [Result] Michel M, Trafton J, Martins S, Wang D, Tu S, Johnson N, Goldstein MK. Improving Patient Safety Using ATHENA-Decision Support System Technology: The Opioid Therapy for Chronic Pain Experience. In: Henriksen K, Battles JB, Keyes MA, Grady ML, editors. Advances in Patient Safety: New Directions and Alternative Approaches (Vol. 4: Technology and Medication Safety). Rockville (MD): Agency for Healthcare Research and Quality (US); 2008 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK43756/ PMID 21249951
- [Result] Bosworth HB, Olsen MK, Dudley T, Orr M, Goldstein MK, Datta SK, McCant F, Gentry P, Simel DL, Oddone EZ. Patient education and provider decision support to control blood pressure in primary care: a cluster randomized trial. Am Heart J. 2009 Mar;157(3):450-6. doi: 10.1016/j.ahj.2008.11.003. Epub 2009 Jan 10. PMID 19249414
- [Result] Goldstein MK. Using health information technology to improve hypertension management. Curr Hypertens Rep. 2008 Jun;10(3):201-7. doi: 10.1007/s11906-008-0038-6. PMID 18765090
- [Result] Cucciare MA, Ketroser N, Wilbourne P, Midboe AM, Cronkite R, Berg-Smith SM, Chardos J. Teaching motivational interviewing to primary care staff in the Veterans Health Administration. J Gen Intern Med. 2012 Aug;27(8):953-61. doi: 10.1007/s11606-012-2016-6. Epub 2012 Feb 28. PMID 22370769
- [Result] Steinman MA, Goldstein MK. When tight blood pressure control is not for everyone: a new model for performance measurement in hypertension. Jt Comm J Qual Patient Saf. 2010 Apr;36(4):164-72. doi: 10.1016/s1553-7250(10)36028-4. PMID 20402373

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study initially involved 5 medical centers with 103 participants across the medical centers. One of the 5 medical centers completed installation of ATHENA-HTN system, but did not continue with the intervention period, so the intervention included 4 medical centers with 82 participants.
Units Other Than Participants: Clinic sites within medical centers
Groups:
- Guideline Link Only: Link to The Seventh Report of the Joint National Committee on Prevention Detection Evaluation and Treatment of High Blood Pressure (JNC7) and to VA-Department of Defense (DoD) hypertension guidelines
  Link to Hypertension Guidelines: Primary care providers were sent, once, a link (URL) to the VA-DoD and JNC7 hypertension guidelines.
- ATHENA-CDS-HTN: ATHENA display providing guideline-based recommendations to clinicians at the time of patient care. Link to JNC7 guidelines.
  ATHENA-Hypertension clinical decision support system: ATHENA display provides guideline-based recommendations to clinicians at the time of patient care.
Period: Overall Study
Arm/Group | Guideline Link Only | ATHENA-CDS-HTN
Started (Randomization of the clinic sites.) | 34; 10 Clinic sites within medical centers | 48; 10 Clinic sites within medical centers
Intervention Started | 30; 10 Clinic sites within medical centers | 46; 10 Clinic sites within medical centers
Completed | 29; 10 Clinic sites within medical centers | 43; 10 Clinic sites within medical centers
Not Completed | 5; 0 Clinic sites within medical centers | 5; 0 Clinic sites within medical centers
Not completed — Left clinic before intervention started | 4 | 1
Not completed — Change in job role before intervention | 0 | 1
Not completed — Left clinic after intervention started | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of primary care providers who started intervention period
Units Other Than Participants: clinics
Groups:
- Guideline Link Only: Link to JNC7 and to VA-DoD hypertension guidelines
  Link to Hypertension Guidelines: Primary care providers were sent, once, a link (URL) to the VA/DoD and JNC7 hypertension guidelines.
- Total: Total of all reporting groups
Arm/Group | Guideline Link Only | ATHENA-CDS-HTN | Total
Number analyzed (Participants) | 30 | 46 | 76
Number analyzed (clinics) | 10 | 10 | 20
Age, Customized [Count of Participants; unit: Participants]
  Age >= 18 years | 30 | 46 | 76
Sex/Gender, Customized [Number; unit: percentage of male participants] — Measured percentage of male participants per clinic site, then mean of these percentages for study arm.
  percentage of male participants
    Mean percentage male participants per clinic | 35.5 | 24.6 | 30.1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 46 | 76

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentages of Events After Index Visit to Primary Care by Patient
Description: The outcome measure was mean percentages of Events after index visit to primary care by patients. The Events were the first event in the patient record after the index clinic visit for the patient, as follows. Event 1 is intensification of pharmacotherapy for hypertension. Event 2 is patient achieves below-target blood pressure (BP). Event 3 is patient does not achieve below-target BP nor is there intensification of pharmacotherapy for hypertension. Event 4 is patient does not achieve BP target, does not have intensified pharmacotherapy, and does not return for further BP measurements. Each patient was assigned one and only one Event. If a patient has pharmacotherapy intensified and also achieved BP below-target, the patient was assigned to whichever happened first. An initial model fitting all 4 events did not detect a difference by study arm for mean percentage of Event 4; final findings are based on a denominator of Events 1 - 3.
Time Frame: up to one year after index visit
Measure: Number; unit: mean percentage of events
Units Other Than Participants: clinic sites
Groups:
- Guideline Link Only: Link to JNC7 and to VA-DoD hypertension guidelines
  Link to Hypertension Guidelines: Primary care providers were sent, once, a link (URL) to the VA/DoD and JNC hypertension guidelines.
Arm/Group | Guideline Link Only | ATHENA-CDS-HTN
Number analyzed (Participants) | 30 | 46
Number analyzed (clinic sites) | 10 | 10
mean percentage of events
  Event 1 | 25.4 | 30.6
  Event 2 | 59.6 | 55.2
  Event 3 | 16.2 | 13.7
Statistical Analysis 1: Comparison: Guideline Link Only vs ATHENA-CDS-HTN; We compared the mean percentages of events per clinician between study arms, using mixed model regression adjusting for medical center, clinic type (community-based clinic vs not), clinician discipline (MD vs non-MD), presence of pharmacist in the clinic, and mean age of clinician's panels of patients as fixed effects, and clinic as a random effect to account for clustering of clinicians within clinics; Test type: Other; p > 0.1, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Up to one year.
Description: The study did not provide any intervention to patients. Patients were receiving their usual care from their primary care providers (clinicians.) The providers in the study were the study participants. The providers were theoretically at risk that the study might identify or disclose adverse information about their clinical management of patients. Another theoretical risk was that a provider might find the clinical decision support intrusive and problematic for clinical care.
Groups:
- Guideline Link Only: Guideline Link Only. Link to JNC7 and to VA-DoD hypertension guidelines
  Guideline Link Only: Primary care providers were sent, once, a link (URL) to the VA/DoD and JNC hypertension guidelines.
- ATHENA-CDS-HTN Plus Guideline Link: ATHENA-Clinical Decision Support (CDS)-HTN plus Guideline Link. ATHENA-CDS-HTN display on the cover sheet of electronic health record, plus link to the guidelines
  ATHENA-CDS-HTN plus Guideline Link: ATHENA-CDS-HTN display provides guideline-based recommendations to clinicians at the time of patient care.
Arm/Group | Guideline Link Only | ATHENA-CDS-HTN Plus Guideline Link
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/46
Other Adverse Events (participants affected / at risk) | 0/31 | 0/46

LIMITATIONS AND CAVEATS:
The study has originally planned to include 5 large medical centers. One of the medical centers dropped out before the intervention started. This lowered the number of clinic sites and of participants (clinicians).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes